CLINICAL TRIAL: NCT05773833
Title: Osage Community Supported Agriculture
Brief Title: Indigenous Supported Agriculture "Go Healthy"
Acronym: ISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Collaborators: University of Oklahoma (Other); Osage Nation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021026
Record Dates: First submitted 2023-02-24; First posted 2023-03-17 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Diet, Healthy; Blood Pressure; Overweight or Obesity; Food Insecurity; Health Status
Keywords: Blood Pressure; Obesity; CBPR; American Indian; BMI; Food Environment; Blood Lipids
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Go Healthy" Intervention Group (Experimental): "Go Healthy" program
  Interventions: Behavioral: "Go Healthy" program
- Wait-list Control Group (No Intervention): Monetary compensation equal in value to the "Go Healthy" program

INTERVENTIONS:
Behavioral: "Go Healthy" program — Weekly food boxes of fresh fruits and vegetables for 16 weeks; healthy eating and traditional foods curriculum available inside the box; monthly in-person healthy eating and traditional Indigenous foods cooking workshop; Indigenous cooking demonstration video website links to accompany recipes; and a kitchen starter kit with kitchen cooking supplies
  Arms: "Go Healthy" Intervention Group

SUMMARY:
Native Americans (NAs) have limited access to healthy food and a high prevalence of diet-related diseases. This study will implement an agricultural and health education program in which NA residents of Osage Nation will receive a weekly share of healthy fresh produce coupled with healthy recipes and cooking materials. The program's effect on diet and health outcomes and it's cost-effectiveness will be evaluated, and study processes and findings will be broadly disseminated to support tribes in improving diet and health.

DETAILED DESCRIPTION:
The study will implement a new community supported agriculture (CSA) program, which the investigators refer to as the "Go Healthy" Indigenous Supported Agriculture (ISA) program, in which citizens in Osage Nation will receive a weekly share of fresh fruits and vegetables for 16 weeks. The investigators will test the efficacy of the "Go Healthy" program combined with culturally-tailored nutrition and cooking education on diet and health outcomes among NA households, evaluate its cost-effectiveness, and develop a multimedia toolkit for disseminating findings.

Specific Aims:

1. Conduct a randomized controlled trial to test the newly developed ISA program's effect on diet, blood pressure, and blood lipids (primary outcomes) and on body mass index (BMI), hemoglobin A1c (HbA1c), food insecurity, health status, and Skin carotenoid measurement by Veggie Meter (secondary outcomes) among 200 NA households (400 adults and up to 400 children) with an index household adult (aged 18-75) identifying as NA with overweight/obesity;
2. Perform an economic evaluation for individual (e.g., health-related quality of life), organizational (e.g., healthcare utilization costs), and community-level (e.g., prevention of cardiometabolic diseases) outcomes; and
3. Document and disseminate study processes and findings using participatory video methods, and compile a web-based toolkit for other NA communities to use to improve tribal food systems

ELIGIBILITY:
Adult Participant Inclusion Criteria:

* 18-75 years of age
* Identify as Native American (index adult participant only)
* Reside in Osage Nation
* Plan to stay in Osage Nation in the next year
* Overweight ot obesity, defined as BMI >= 25 kg/m2, measured by research staff (index adult participant only)
* Willing and able to follow study procedures

Child Participant Inclusion Criteria:

* 3-17 years of age
* Reside in Osage Nation
* Plan to stay in Osage Nation in the next year
* Willing and able to follow study procedures

Exclusion Criteria:

* Those that are pregnant or planning to become pregnant during the study period

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Diet using Healthy Eating Index scores | Measured at baseline and immediately post-intervention (16 weeks)
  Change in vegetable and fruit intake using the National Cancer Institute's Automated Self-Administered 24-hour Recall (ASA-24) 2022. This self-report instrument generates a "healthy eating index" (HEI), with scores ranging from 0 (least healthy) to 100 (healthiest). Continuous values of the overall HEI score will constitute our primary outcome.
Blood pressure (adults only) | Measured at baseline and immediately post-intervention (16 weeks)
  Change in systolic and diastolic blood pressure
HDL (adults only) | Measured at baseline and immediately post-intervention (16 weeks)
  Change in HDL levels measured in mg/dL
LDL (adults only) | Measured at baseline and immediately post-intervention (16 weeks)
  Change in LDL levels measured in mg/dL
Total cholesterol (adults only) | Measured at baseline and immediately post-intervention (16 weeks)
  Change in total cholesterol levels measured in mg/dL
Glucose (adults only) | Measured at baseline and immediately post-intervention (16 weeks)
  Change in glucose levels measured in mg/dL
Triglycerides (adults only) | Measured at baseline and immediately post-intervention (16 weeks)
  Change in triglyceride levels measured in mg/dL

SECONDARY OUTCOMES:
BMI status using CDC guidelines | Measured at baseline and immediately post-intervention (16 weeks)
  Change in BMI will be calculated by dividing weight in kilograms by height in meters squared. Using CDC guidelines, adults will be categorized into the following groups based 1) underweight (BMI < 18.5); 2) healthy weight (BMI = 18.5-24.9); 3) overweight (BMI = 25.0-29.9); 4) obese (BMI = 30.0-39.9), and 5) morbidly obese (BMI ≥ 40.0). Child BMI will be calculated as a continuous variable using the CDC Child and Teen BMI Calculator.
HbA1c (adults only) | Measured at baseline and immediately post-intervention (16 weeks)
  Change in HbA1c levels
Food insecurity using the United States Department of Agriculture's Household Food Security Survey Module | Measured at baseline and immediately post-intervention (16 weeks)
  Change in food insecurity using the Household Food Security Module. This instrument contains 18 items to capture the qualitative and quantitative dimensions of household food supply, including psychological and behavioral responses of household members. To compute levels of food security and insecurity, we will total the number of affirmative responses to these items, counting "Often" and "Sometimes" as affirmative. Consistent with USDA guidelines, 0-2 affirmatives indicate food security, and 3 or more affirmatives indicate food insecurity.
Overall health status using the Short Form-36 | Measured at baseline and immediately post-intervention (16 weeks)
  Change in overall health status with answer options of excellent, very good, good, fair, or poor using the Short Form-36.
Skin Carotenoids | Measured at baseline and immediately post-intervention (16 weeks)
  Change in skin carotenoid score using the Veggie Meter instrument (scale ranging from 0 to 800). Higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Valarie Jernigan, DrPH, Principal Investigator — Oklahoma State University Center for Health Sciences
Locations (1):
- The Osage Nation, Pawhuska, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No